CLINICAL TRIAL: NCT04353466
Title: An Open-label, Investigator Initiated Clinical Trial to Asses Impact of Elelyso on Bone Involvement in Patients With Gaucher Disease Currently Treated With Other ERTs
Brief Title: Assessing the Impact of Elelyso on Bone Involvement Currently Treated With Other ERTs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Ari Zimran, Prof., Shaare Zedek Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 138-16-SZMC
Record Dates: First submitted 2020-04-13; First posted 2020-04-20 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Gaucher Disease, Type 1
MeSH Terms: conditions — Gaucher Disease | interventions — taliglucerase alfa

STUDY DESIGN:
Intervention Model Description: The objective of this study is to assess Elelyso treatment on bone disease in Gaucher patients currently treated with other enzyme replacement therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Trial to asses impact of Elelyso on bone involvement in patien (Experimental): The infusions will be administered at the selected medical center or in the home care setup. The dose of intravenous (IV) infusions of Elelyso will be the same dose of the other ERTs . Bone parameters QCSI and BMD will be assessed at baseline, 12 months and 24 months.
  Interventions: Procedure: quantitative chemical shift imaging (QCSI); Drug: Elelyso

INTERVENTIONS:
Procedure: quantitative chemical shift imaging (QCSI) — Poor scores of QCSI with Fat Fraction below the cut off point of 0.3 which is considered "bone at risk"
Drug: Elelyso — intravenous (IV) infusions of Elelyso
  Other Names: Taliglucerase Alfa

SUMMARY:
The objective of this study is to assess Elelyso treatment on bone disease in Gaucher patients currently treated with other enzyme replacement therapy.

Experience from early access program (2009-2012) has suggested that some patients who have been stable on imiglucerase have shown poor scores of QCSI with Fat Fraction below the cut off point of 0.23 which is considered "bone at risk", and have demonstrated remarkable improvement upon switching to Elelyso, including particularly 2 patients who did not have any change in dose or any drug interruption prior to the switch.

These findings may be explained by the better glycan structure of imiglucerase (see Tekoah et al, 2013). The fact that in many patients prevention of bony complications is the main indication for ERT highlights the importance of this study, as all clinical trials of all ERTS heretofore did not include the bones as primary or secondary end-points but only as exploratory, and as such had only limited value,

DETAILED DESCRIPTION:
Open-label study in patients with Gaucher disease currently treated with commercial ERTs. Eligible patients will receive intravenous (IV) infusions of Elelyso every two weeks. The infusions will be administered at the selected medical center or in the home care setup. The dose of Elelyso will be the same dose of the other ERTs . Bone parameters QCSI and BMD will be assessed at baseline, 12 months and 24 months.

The intention is to open 3 more sites in Israel thereby making this IIR a multi center national trial

ELIGIBILITY:
Inclusion Criteria:

* GD patients, male and female, 18 years or older
* Currently treated with enzyme replacement therapy for 5 years and more, with a stable unchanged dose in the previous 6 months
* Imaging features of significant residual bone disease defined as QCSI under 0.3 bone at risk
* Able to provide written informed consent

Exclusion Criteria:

* Currently taking another experimental drug for any condition
* Presence of any medical, emotional, behavioral or psychological condition that in the judgment of the Investigator would interfere with the patient's compliance with the requirements of the study.
* Past exposure to Elelyso

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
QCSI results at 12 months, Fat fraction under 0.3. | 12 months
  Improvement of QCSI results in patients with Gaucher disease currently treated with commercial ERTs. Eligible patients will receive intravenous (IV) infusions of Elelyso every two weeks. The infusions will be administered at the selected medical center or in the home care setup. The dose of Elelyso will be the same dose of the other ERTs . Bone parameters QCSI and BMD will be assessed at 12 months.
QCSI results at 24 months, Fat fraction under 0.3. | 24 months
  Improvement of QCSI results in patients with Gaucher disease currently treated with commercial ERTs. Eligible patients will receive intravenous (IV) infusions of Elelyso every two weeks. The infusions will be administered at the selected medical center or in the home care setup. The dose of Elelyso will be the same dose of the other ERTs . Bone parameters QCSI and BMD will be assessed at 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ari Zimran, MD, Principal Investigator — Shaheed Ziaur Rahman Medical College

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] van Dussen L, Zimran A, Akkerman EM, Aerts JM, Petakov M, Elstein D, Rosenbaum H, Aviezer D, Brill-Almon E, Chertkoff R, Maas M, Hollak CE. Taliglucerase alfa leads to favorable bone marrow responses in patients with type I Gaucher disease. Blood Cells Mol Dis. 2013 Mar;50(3):206-11. doi: 10.1016/j.bcmd.2012.11.001. Epub 2012 Nov 28. PMID 23199589
- [Result] Zimran A, Dinur T, Revel-Vilk S, Akkerman EM, van Dussen L, Hollak CEM, Maayan H, Altarescu G, Chertkoff R, Maas M. Improvement in bone marrow infiltration in patients with type I Gaucher disease treated with taliglucerase alfa. J Inherit Metab Dis. 2018 Nov;41(6):1259-1265. doi: 10.1007/s10545-018-0195-y. Epub 2018 Jul 31. PMID 30066229
- [Result] van Dussen L, Akkerman EM, Hollak CE, Nederveen AJ, Maas M. Evaluation of an imaging biomarker, Dixon quantitative chemical shift imaging, in Gaucher disease: lessons learned. J Inherit Metab Dis. 2014 Nov;37(6):1003-11. doi: 10.1007/s10545-014-9726-3. Epub 2014 Jun 13. PMID 24924293